CLINICAL TRIAL: NCT02198612
Title: FREEDOM: "Pilot Study of the Feasibility and Safety of Resuming Early Walking After Manual Compression in Patients Treated for Peripheral Artery Disease by Endovascular Technique Involving Retrograde Femoral Puncture"
Acronym: FREEDOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RC14_0226
Record Dates: First submitted 2014-07-15; First posted 2014-07-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manual puncture point compression (Other): Manual puncture point compression following a diagnostic or therapeutic procedure by endovascular technique involving retrograde femoral puncture point with 5F guide catheter
  Interventions: Other: Manual puncture point compression

INTERVENTIONS:
Other: Manual puncture point compression — Manual puncture point compression following a diagnostic or therapeutic procedure by endovascular technique involving retrograde femoral puncture point with 5F guide catheter

SUMMARY:
Over the past years, arterial closure systems have tended to replace manual compression to ensure hemostasis at femoral artery puncture points. Arterial closure systems reduce hemostasis and patient immobilization times, thus enabling early resumption of walking. These devices have contributed extensively to the development of outpatient stays for cardiology, vascular and neuro-radiology procedures.

According to certain studies however, it would appear that arterial closure devices do not present any greater benefits than manual compression in terms of hemostasis and complications. Moreover, the use of increasingly small diameter instruments would tend to render manual compression sufficient. Finally, the use of these devices generates additional costs.

The purpose of our study is to evaluate the feasibility and safety of manual compression before early resumption of walking in patients managed by conventional hospitalization for a diagnostic or therapeutic endovascular procedures by retrograde femoral puncture with 5F guide catheter.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Endovascular examination or treatment compatible with a 5F guide catheter
* Walking ability
* Patient affiliated with a social security scheme
* Patient's signed informed consent form

Exclusion Criteria:

* Underage patient
* Patient of age, but under legal guardianship or care
* Contraindication to endovascular treatment
* Use of a 6F or greater guide catheter
* Morbidity contraindicating same-day walking
* History of punctured open femoral triangle surgery
* Radial or humeral puncture
* Bilateral femoral puncture
* Anterograde femoral puncture
* Acute ischemia
* Anticoagulant treatment
* Allergy to Elastoplast® type adhesive strips
* Life expectancy of less than one month
* Patient refusal to take part in the study
* Participation in another therapeutic trial
* Pregnant woman
* Patients who do not speak French, refusing or incapable of the follow-up proposed by the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Resumption of walking at H5 will be evaluated by a walking test | Hour 5
  To demonstrate the feasibility of early resumption of walking after manual puncture point compression following a diagnostic or therapeutic procedure by endovascular technique involving retrograde femoral puncture point with 5F guide catheter.

SECONDARY OUTCOMES:
Occurrence of major punctured femoral triangle events during the perioperative period, requiring prolongation of hospitalization, repeat hospitalization or repeat surgery (hematoma, hemorrhage or false aneurysm) | Hour 5
Occurrence of minor punctured femoral triangle events during the perioperative period, not requiring prolongation of hospitalization, repeat hospitalization or repeat surgery | Hour 5
Time to onset of complications | Hour 5
Puncture point pain (visual analog scale of pain) | Hour 5
Quality of life evaluation (EQ5D questionnaire) | Month 1
Compression time | Hour 5

CONTACTS AND LOCATIONS:
Overall Officials: Yann GOUEFFIC, Professor, Study Chair — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France